CLINICAL TRIAL: NCT05551429
Title: Factors Associated With Participation in Hospital-Based Cardiac Rehabilitation Program in Patients With Acute Coronary Syndrome
Brief Title: Factors Related to Participation in Cardiac Rehabilitation in Patients With Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Levent Karataş, Principal Investigator, Gazi University
Other Study IDs: Participation in Cardiac Rehab
Record Dates: First submitted 2022-09-15; First posted 2022-09-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Acute Coronary Syndrome; Cardiovascular Diseases; Cardiac Rehabilitation
Keywords: Acute Coronary Syndrome; Cardiac Rehabilitation; Myocardial Infarction; Participation; Health Literacy; Rehabilitation Barriers
MeSH Terms: conditions — Acute Coronary Syndrome; Cardiovascular Diseases; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Acute Coronary Syndrome: The study sample will comprise acute coronary syndrome patients admitted to Gazi University Faculty of Medicine, Cardiology Department, Coronary Intensive Care Unit because of one or more of the diagnoses of acute ST-elevation myocardial infarction (MI), acute non-ST elevation MI and unstable angina pectoris. Patients who are hemodynamically stable and have no signs of residual ischemia after acute care will be informed by the cardiologist about the study. After the inclusion process, patients will be evaluated in terms of clinical characteristics, muscle strength, quality of life, and health literacy. They will be given detailed information about CR and an appointment will be made four weeks later for starting the exercise program. In the follow-up, the Cardiac Rehabilitation Barriers Scale-Turkish Version will be applied to those who do not participate in the initial exercise program.
  Interventions: Behavioral: Invitation to the CR

INTERVENTIONS:
Behavioral: Invitation to the CR — 1. Oral and written information emphasise the benefits of cardiac rehabilitation in terms of treatment of heart diseases, increasing functional capacity, reducing morbidity and mortality, and enhancing secondary prevention.
  2. Introducing the scope and method of administration of CR to patients.
  3. Setting up the appointment for the initial CR session four weeks later.

SUMMARY:
Acute coronary syndrome (ACS) is one of the most important causes of mortality and morbidity all over the world. Cardiac rehabilitation (CR) is a crucial part of secondary prevention and optimal care of patients with ACS. However, the participation rate in CR after ACS is far from expected. In our study, we will aim to examine the rate of participation in cardiac rehabilitation and the factors affecting it in patients followed up for acute coronary syndrome in the coronary intensive care unit of our hospital. Our main hypothesis is that the lower rate of participation in cardiac rehabilitation in patients with acute coronary syndrome is associated with one or more of that older age, female gender, multimorbidity, poor functional capacity, lower health literacy level or quality of life levels.

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) is an umbrella term comprising unstable angina, myocardial infarction (MI) with or without ST-segment elevation, and sudden cardiac death because of acute myocardial ischemia. ACS is one of the most important causes of mortality and morbidity all over the world. Today, cardiac rehabilitation has become an integral part of the medical care and secondary prevention programs of cardiovascular diseases including ACS. Cardiac rehabilitation (CR) is a long-term comprehensive rehabilitation program that includes but not limited to patient evaluation, determination of risk profile, patient-tailored exercise training, and behavioural and lifestyle changes aiming at risk reduction in cooperation with many disciplines. It consists of comprehensive interventions. Despite its known benefits and recommended in national and international guidelines, the participation rate in cardiac rehabilitation is lower than expected. Studies involving different countries and societies showed that lower participation was associated with inadequate referral, female gender, poor motivation, older age, comorbidities, difficulty in transportation, and poor socioeconomic status. It has been suggested that setting up a CR appointment before discharge via clinical visits by the CR team or automatic referral systems, increasing patient interest and knowledge through written invitations and brochures, and providing support for transportation may increase participation in CR.

In our country, there are not enough studies addressing the success of participation and compliance in cardiac rehabilitation. In this study, we aim to determine patient related factors associated with low participation in CR in patients admitted to our coronary intensive care unit (ICU) with ACS diagnosis. All patients included in this study will be comprehensively informed about CR and the initial CR session will be scheduled to minimize effect of inadequate referral.

ELIGIBILITY:
Inclusion Criteria:

* Being hospitalized in the coronary intensive care unit with the diagnosis of acute coronary syndrome
* Being able to walk and get up from a chair without the support of a person
* Agree to take part in the study

Exclusion Criteria:

* Presence of any conditions that prevent exercise training (severe orthopaedic, neurological or rheumatological disease, acute infection, acute pericarditis, endocrine and metabolic disorders, etc.)
* Presence of neuropsychiatric diseases or conditions that may prevent cooperation
* Persisting unstable angina
* Having severe stenosis or insufficiency of heart valve
* Congenital structural heart diseases
* Presence of decompensated heart failure
* Uncontrolled arrhythmias that may cause hemodynamic instability during exercise
* Exercise contraindication decision of the cardiologist

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-75 years admitted to the coronary intensive care unit with the diagnosis of acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Rate of participation in the CR | Four weeks after discharge from ICU
  Number of patients admitted to the first CR session four weeks after discharge from the ICU

SECONDARY OUTCOMES:
Timed Up and Go Test | At initial evaluation of the participant in ICU
  It is a test that evaluates balance, mobility and lower extremity muscle strength, which includes getting up from a chair, walking 3 meters, turning back and sitting on the chair again. After an adaptation trial, the test is performed twice, including a rest period between trials. Patients are allowed to use any assistive device such as a cane or walker. The main result is the average duration of the two trials. A longer test time indicates worse performance.
Measurement of hand grip strength | At initial evaluation of the participant in ICU
  Hand grip strength is an important indicator of overall muscle strength. Measurements will be performed using a Jamar dynamometer, while sitting, with the arm just next to the trunk, the elbow flexed to 90 degrees, and the forearm and wrist in a neutral position, as recommended by the American Association of Hand Therapists. Three measurements will be performed, including one-minute intervals between trials. The highest result of the three trials will be accepted.
Two minute Step Test | At initial evaluation of the participant in ICU
  This test is used to evaluate the endurance of lower extremity muscles. The patient is asked to stand next to a wall. The midpoint of the distance between the patient's iliac crest and the knee is measured and marked on the wall. On the signal "go" the patient begins stepping (not running) in place, raising each knee to the mark on the wall, as many times as possible in the 2 minutes. The number of times the right knee reaches the required height is counted. If the proper knee height cannot be maintained, the patient is asked to slow down or to stop until he/she can regain the proper form, while keeping the stopwatch running.
World Health Organization Quality of Life Scale-Short Form | At initial evaluation of the participant in ICU
  This scale is used for a brief assessment of the quality of life in routine clinical practice, large-scale epidemiological studies, or clinical trials. It comprises 27 questions that evaluate general health status, physical health, psychological status, social relations and environmental issues sub-titles. Each question receives an answer corresponding to 1-5 points. The percentages of the scores obtained from each sub-title allow us to make a quantitative interpretation of domains of the quality of life.
Turkish Health Literacy Scale-32 | At initial evaluation of the participant in ICU
  Turkish Health Literacy Scale-32 ("Türk Sağlık Okuryazarlık Ölçeği" in Turkish) is a survey comprising 32 questions that measure health literacy. It is derived from the Turkish version of The European Health Literacy Survey, which consists of 47 questions. It has been reported to be valid and reliable in Turkish population.
  The survey addresses accessing, understanding, evaluating and using/applying health-related information. Each question is answered by choosing one of the options "very easy", "easy", "difficult" "very difficult" or "I don't know", corresponding to 4, 3, 2, 1 and null points, respectively. The mean score is calculated after excluding questions with invalid or "I don't know" answers. The index is determined following the formula "index = (mean score - 1) x (50/3)" A score of 0-25 indicates insufficient, >25 to 33 indicates limited, >33 to 42 indicates adequate, and >42 to 50 indicates excellent health literacy.
Cardiac Rehabilitation Barriers Scale-Turkish Version | Four weeks after discharge from ICU
  It is a questionnaire that aims to determine the reason(s) for not attending or missing the CR sessions. Each of the 21 possible reasons is answered by the patient on a 1-5 Likert scale (strongly disagree-disagree-decided-agree-strongly disagree). The last question has an open-ended answer option for patient to report other reasons. Turkish version of this survey were found to be valid and reliable by Coşkun et al. in 2019.
  Patients who do not attend to their CR appointment at fourth week after discharge will be called and the Cardiac Rehabilitation Barriers Scale-Turkish Version will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Nesrin Demirsoy, MD, Principal Investigator — Gazi University Faculty of Medicine; Levent Karataş, MD, Principal Investigator — Gazi University Faculty of Medicine
Locations (1):
- Gazi University Hospital, Department of Physical Medicine and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Price KJ, Gordon BA, Bird SR, Benson AC. A review of guidelines for cardiac rehabilitation exercise programmes: Is there an international consensus? Eur J Prev Cardiol. 2016 Nov;23(16):1715-1733. doi: 10.1177/2047487316657669. Epub 2016 Jun 27. PMID 27353128
- [Background] Pio CSA, Chaves G, Davies P, Taylor R, Grace S. Interventions to Promote Patient Utilization of Cardiac Rehabilitation: Cochrane Systematic Review and Meta-Analysis. J Clin Med. 2019 Feb 5;8(2):189. doi: 10.3390/jcm8020189. PMID 30764517
- [Background] Grace SL, Krepostman S, Brooks D, Jaglal S, Abramson BL, Scholey P, Suskin N, Arthur H, Stewart DE. Referral to and discharge from cardiac rehabilitation: key informant views on continuity of care. J Eval Clin Pract. 2006 Apr;12(2):155-63. doi: 10.1111/j.1365-2753.2006.00528.x. PMID 16579824
- [Background] Ades PA, Keteyian SJ, Wright JS, Hamm LF, Lui K, Newlin K, Shepard DS, Thomas RJ. Increasing Cardiac Rehabilitation Participation From 20% to 70%: A Road Map From the Million Hearts Cardiac Rehabilitation Collaborative. Mayo Clin Proc. 2017 Feb;92(2):234-242. doi: 10.1016/j.mayocp.2016.10.014. Epub 2016 Nov 15. PMID 27855953
- [Background] Coşkun, Özge Keniş, et al. Validity and reliability of the Turkish version of cardiac rehabilitation barriers scale. Gülhane Tip Dergisi 61.2 (2019): 59.
- [Background] Okyay, P., et al. A new Health Literacy Scale: Turkish Health Literacy Scale and its psychometric properties: Pinar Okyay. The European Journal of Public Health 25.suppl_3 (2015): ckv175-220.
- See also: WHO methods and data sources for country-level causes of death 2000-2019 — http://www.who.int/docs/default-source/gho-documents/global-health-estimates/ghe2019_cod_methods.pdf
- See also: Turkish Health Literacy Survey (TSOY-32) — https://ekutuphane.saglik.gov.tr/Home/GetDocument/530